CLINICAL TRIAL: NCT07096258
Title: A Patient Registry Collecting the Clinical and Molecular Profiling Data of Patients With Locally Advanced and/or Metastatic, Unresectable, Stages IIIB/C or IV Non-small Cell Lung Cancer (NSCLC), Who Have Not Previously Been Treated for This Advanced Disease and Are Therefore Considered as Patients Receiving First-line Therapy.
Brief Title: EMPATHY NSCLC: European Registry for Plasma-Based Molecular Profiling in Advanced NSCLC Patients
Acronym: EMPATHY NSCLC
Status: Recruiting | Type: Observational
Sponsor: Hedera Dx SA (Industry)
Responsible Party: Sponsor
Other Study IDs: EMPATHY NSCLC
Record Dates: First submitted 2025-07-24; First posted 2025-07-31 (Actual); Last update posted 2025-07-31 (Actual); Status verified 2025-07

CONDITIONS: NSCLC (Advanced Non-small Cell Lung Cancer)
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Advanced NSCLC patients

SUMMARY:
The goal of this registry is to capture real-world data from plasma- and tissue-based molecular profiling, treatments, outcomes and patient-reported outcomes from patients with advanced or metastatic non-small cell lung cancer (NSCLC). The main objective of the study is to better understand the real-world clinical practice of the use and utility of molecular tumour profiling, the choice of treatment, and the outcome after such molecular profiling and treatment.

ELIGIBILITY:
Inclusion Criteria:

* Locally advanced or metastatic, unresectable NSCLC, stages IIIB/C or IV, who have not previously been treated for this advanced disease.
* Intention-to-initiate first-line tumour therapy for this advanced disease.
* Eastern Cooperative Oncology Group (ECOG) performance status ≤ 2.
* At least 18 years of age on the day of signing informed consent, and capable of signing informed consent.

Exclusion Criteria:

* Any known non-cutaneous malignancy (except for this NSCLC and early-stage non-invasive cervical cancer) that has occurred within 5 years prior to enrolment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Cancer Hospitals
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2024-06-01 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2031-12 (Estimated)

PRIMARY OUTCOMES:
Actionable biomarkers | At baseline
  Proportion of patients with successful molecular profiling and detectable actionable biomarkers

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Christian Meisel, MD PhD, Study Director — Hedera Dx
Locations (4):
- Université de Lorraine, Nancy, Lorraine, France
- University of Naples "Federico II", Napoli, Italy
- General Universitario Gregorio Marañon, Madrid, Spain
- Hôpitaux Universitaires Genève, Geneva, Canton of Geneva, Switzerland

IPD SHARING:
Plan to Share IPD: Yes
Clinical investigators may request appropriate access to individual de-identified data via the EMPATHY NSCLC Steering Committee.